CLINICAL TRIAL: NCT03030807
Title: Recognition of Pulmonary Hypertension in Patients With Hypersensitivity Pneumonitis
Brief Title: Pulmonary Hypertension in Hypersensitivity Pneumonitis
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Institute for Lung Vascular Research (Other)
Responsible Party: Sponsor
Other Study IDs: 28-037 ex 15/16
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: Right heart catheterization (in case of suspected PH)

SUMMARY:
The investigation serves the identification of pulmonary hypertension (PH) among patients with hypersensitivity pneumonitis (HP). The exact prevalence of PH in HP is unknown. Data from South America indicate that the prevalence of pre-capillary PH amongst patients with HP is higher than 20%. There are no reliable data from Europe so far. According to the investigators previous analysis, more than 400 HP patients have participated in pulmonary rehabilitation at least once in the past 10 years at Klinikum Bad Gleichenberg (Rehabilitation Center for Agricultural Workers in Austria). This collective of patients is to be invited to participate in the study.

A diagnostic algorithm will be applied in the clinical trial, in the case of clinical suspicion the diagnosis of PH will be confirmed by right heart catheterization. Besides the determination of the prevalence of PH in patients with HP the investigators aim to assess the reliability of non-invasive methods (e.g. Echocardiography, ECG...) to predict PH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Hypersensitivity Pneumonitis
* written consent
* Age: 18-90 years

Exclusion Criteria:

* severe impairment of the general health condition
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed Hypersensitivity Pneumonitis
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of pulmonary hypertension | 4 year

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz